CLINICAL TRIAL: NCT06738485
Title: A Phase 3, Open-label, Multicenter, Pharmacokinetics, Efficacy, and Safety Study of a Recombinant Single-chain Factor VIII (rVIII-SingleChain) in Chinese Previously Treated Patients (PTPs) With Hemophilia A
Brief Title: Recombinant Single-chain Factor VIII (rVIII-SingleChain) in Chinese Participants With Hemophilia A Previously Treated With FVIII Products
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CSL627_3003; 2023-001026-34 (EudraCT Number)
Record Dates: First submitted 2024-12-12; First posted 2024-12-17 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Congenital Hemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- rVIII-SingleChain (Experimental): Participants will receive rVIII-SingleChain as an intravenous (IV) infusion for a minimum of 50 exposure days (EDs).
  Interventions: Biological: Recombinant single-chain factor VIII (rVIII-SingleChain)

INTERVENTIONS:
Biological: Recombinant single-chain factor VIII (rVIII-SingleChain) — Lyophilized powder for solution for intravenous injection
  Other Names: CSL627

SUMMARY:
For bridging the available global clinical data of rVIII-SingleChain, with the Chinese population, the aim of this study in China is to investigate the pharmacokinetics (PK) of rVIII-SingleChain after an initial and repeat dose and to assess efficacy and safety during 2 to 3 times weekly prophylaxis treatment with rVIII-SingleChain in male Chinese PTPs with severe hemophilia A (FVIII activity less than [<] 1%).

ELIGIBILITY:
Inclusion Criteria:

* • Male Chinese participants <= 65 years of age.
* • Participants with severe hemophilia A (FVIII activity < 1%).
* • Participants who have received FVIII products for >= 150 EDs (>= 6 years of age) or >= 50 EDs (< 6 years of age).

Exclusion Criteria:

* • Known hypersensitivity (allergic reaction or anaphylaxis) to any FVIII product or hamster protein.
* • Known congenital or acquired coagulation disorder other than congenital FVIII deficiency.
* • Currently receiving intravenous (IV) immunomodulating agents such as immunoglobulin or chronic systemic corticosteroid treatment.
* • Receiving any cryoprecipitate, whole blood, or plasma within 30 days before administration of rVIII-SingleChain.
* • Use of traditional or herbal Chinese medicine(s) with an impact on hemophilia, including coagulation, within 28 days before Day 1 and / or refusal to abstain from these during the study until the end of the participant's participation in the study.

Ages: 0 Days to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-09 (Actual); Primary Completion 2026-06-26 (Estimated); Study Completion 2026-06-26 (Estimated)

PRIMARY OUTCOMES:
Incremental Recovery (IR) of rVIII-SingleChain | Before, and at 30 minutes after the end of, rVIII-SingleChain administration on Day 1
Maximum Concentration (Cmax) of rVIII-SingleChain | Before, and up to 72 hours (participants ≥ 12 years ) and 48 hours (participants < 12 years) after rVIII-SingleChain administration on Day 1
Area Under the Plasma Concentration Time Curve from Time Zero to the Last Measurable Concentration (AUC0-last) of rVIII-SingleChain | Before, and up to 72 hours (participants ≥ 12 years ) and 48 hours (participants < 12 years) after rVIII-SingleChain administration on Day 1
Area Under the Plasma Concentration Time Curve from Time Zero to Infinity (AUC0-inf) of rVIII-SingleChain | Before, and up to 72 hours (participants ≥ 12 years ) and 48 hours (participants < 12 years) after rVIII-SingleChain administration on Day 1
Half-life (t1/2) of rVIII-SingleChain | Before, and up to 72 hours (participants ≥ 12 years ) and 48 hours (participants < 12 years) after rVIII-SingleChain administration on Day 1
Clearance (Cl) of rVIII-SingleChain | Before, and up to 72 hours (participants ≥ 12 years ) and 48 hours (participants < 12 years) after rVIII-SingleChain administration on Day 1
Annualized Spontaneous Bleeding Rate (AsBR) | Up to 29 weeks after rVIII-SingleChain administration
  AsBR for treated bleeding episodes
Number of participants who develop FVIII inhibitors | During routine rVIII-SingleChain prophylaxis dosing, up to 29 weeks after rVIII-SingleChain administration.

SECONDARY OUTCOMES:
Time to reach maximum concentration (Tmax) of rVIII-SingleChain | Before, and up to 72 hours (participants ≥ 12 years ) and 48 hours (participants < 12 years) after rVIII-SingleChain administration on Day 1
Last Concentration (Clast) of rVIII-SingleChain | Before, and up to 72 hours (participants ≥ 12 years ) and 48 hours (participants < 12 years) after rVIII-SingleChain administration on Day 1
  Last observed quantifiable plasma concentration
IR (participants ≥ 12 years of age) of rVIII-SingleChain (Repeat pharmacokinetic [PK]) | Before, and at up to 72 hours after the end of, rVIII-SingleChain infusion at Week 28
Cmax (participants ≥ 12 years of age) of rVIII-SingleChain (Repeat PK) | Before, and at up to 72 hours after the end of, rVIII-SingleChain infusion at Week 28
AUC0-last of rVIII-SingleChain (Repeat PK) | Before, and at up to 72 hours after the end of, rVIII-SingleChain infusion at Week 28
AUC0-inf of rVIII-SingleChain (Repeat PK) | Before, and at up to 72 hours after the end of, rVIII-SingleChain infusion at Week 28
t1/2 of rVIII-SingleChain (participants ≥ 12 years of age) (Repeat PK) | Before, and at up to 72 hours after the end of, rVIII-SingleChain infusion at Week 28
Cl of rVIII-SingleChain (participants ≥ 12 years of age) (Repeat PK) | Before, and at up to 72 hours after the end of, rVIII-SingleChain infusion at Week 28
Annualized Bleeding Rate (ABR) | Up to 29 weeks after rVIII-SingleChain administration
  Total ABR for treated, untreated, and both treated and untreated bleeding episodes (spontaneous, traumatic, and unknown cause)
Hemostatic Efficacy for Major and Nonmajor Bleeding Episodes | Up to 29 weeks after rVIII-SingleChain administration
  The investigator will rate the efficacy of the rVIII-SingleChain treatment for major and nonmajor bleeding episodes based on a hemostatic efficacy four point rating scale of "excellent, good, moderate or no efficacy".
Consumption of rVIII-SingleChain - number of infusions (doses) | Up to 29 weeks after rVIII-SingleChain administration
Consumption of rVIII-SingleChain - IU/kg per participant per month | Up to 29 weeks after rVIII-SingleChain administration
  rVIII-SingleChain consumption (IU/kg) per participant per month, for the weekly regimen, on-demand treatment, and total treatment.
Consumption of rVIII-SingleChain - IU/kg per participant per year | Up to 29 weeks after rVIII-SingleChain administration
  rVIII-SingleChain consumption (IU/kg) per participant per year, for the weekly regimen, on-demand treatment, and total treatment.
Number of bleeding episodes requiring rVIII-SingleChain to achieve hemostasis | Up to 29 weeks after rVIII-SingleChain administration
  Number of bleeding episodes requiring 1, <= 2, or > 2 infusions (doses) of rVIII-SingleChain to achieve hemostasis
Percentage of bleeding episodes requiring rVIII-SingleChain to achieve hemostasis | Up to 29 weeks after rVIII-SingleChain administration
  Percentage of bleeding episodes requiring 1, <= 2, or > 2 infusions (doses) of rVIII-SingleChain to achieve hemostasis
Number of participants who develop noninhibitory antibodies against rVIII-SingleChain | Before, and up to 29 weeks after, rVIII-SingleChain administration
Number of participants who develop antibodies against Chinese hamster ovary host cell protein | Before, and up to 29 weeks after, rVIII-SingleChain administration
Number of participants with Treatment-emergent Adverse Events (TEAEs), including related TEAEs, and serious adverse events (SAEs) | Up to 33 weeks after rVIII-SingleChain administration
Percentage of participants with TEAEs, including related TEAEs, and serious adverse events (SAEs) | Up to 33 weeks after rVIII-SingleChain administration
Number of TEAEs (events) | Up to 33 weeks after rVIII-SingleChain administration

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — CSL Behring
Locations (20):
- China (20):
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Children's Hospital, Beijing, Beijing Municipality
  - Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Guangzhou Women and Children's Medical Center, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Liuzhou People's Hospital, Liuchow, Guangxi
  - North China University of Science and Technology Affiliated Hospital, Tangshan, Hebei
  - Hospital of Hematology, Chinese Academy of Medical Sciences, Tianjin, Hebei
  - Henan children's hospital Zhengzhou children's Hospital, Zhengzhou, Henan
  - Hunan Provincial Children's Hospital, Changsha, Hunan
  - Nanjing Children's Hospital, Nanjing, Jiangsu
  - XuZhou Children's Hospital, Xuzhou, Jiangsu
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - Quinghai Provincial People's Hospital, Xining, Qinghai
  - Jinan Central Hospital, Jinan, Shandong
  - Qingdao Women and Children's Hospital, Qingdao, Shandong
  - Shanghai Jiaotong University School of Medicine, Ruijin Hospital, Shanghai, Shanghai Municipality
  - The second affiliated hospital of Kunming Medical University, Kunming, Yunan
  - The Children's Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
CSL will consider on a case-by-case basis requests to share Individual Patient Data (IPD) with external bona-fide, qualified scientific and medical researchers. For information on the process and requirements for submitting a voluntary data sharing request for IPD, please contact CSL at clinicaltrials@cslbehring.com.
Supporting Information: Study Protocol, SAP
Time Frame: Requests for IPD will generally be considered once review by major regulatory authorities (i.e., FDA, EMA) is complete and the primary publication is available.
Access Criteria: Proposed research should seek to answer a previously unanswered important medical or scientific question.
  Applicable country specific privacy and other laws and regulations will be considered and may prevent sharing of IPD.
  If the request is approved and the researcher has executed an appropriate data sharing agreement, IPD that has been appropriately anonymized will be available.